CLINICAL TRIAL: NCT06469060
Title: Tislelizumab Combined With Chemotherapy as Neoadjuvant Regimen for AdenoCarcinoma of the Esophagogastric Junction: a Single-arm, Phase II Clinical Trial (TRACE)
Brief Title: Neoadjuvant Immunochemotherapy for Adenocarcinoma of the Esophagogastric Junction
Acronym: TRACE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief of Department of Thoracic Surgery, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCE2403
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: Adenocarcinoma; Esophagogastric Junction; Immunochemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant anti-PD-1 with DOC chemotherapy (Experimental): Drug: Immuno-chemotherapy. Patients will receive neoadjuvant therapy (one cycle of Tislelizumab monotherapy followed by four cycles of Tislelizumab plus Docetaxel, Oxaliplatin and Capecitabine) followed by the esophagectomy.
  Interventions: Drug: neoadjuvant anti-PD-1 with DOC chemotherapy

INTERVENTIONS:
Drug: neoadjuvant anti-PD-1 with DOC chemotherapy — Patients were treated with one cycle of Tislelizumab 200 mg monotherapy on day
  1. At 3 weeks and with intervals of 3 weeks between each cycle (weeks 3, 6, 9 and 12), patients received a total of four combination cycles consisting of Tislelizumab 200 mg, docetaxel 50 mg m-2 and oxaliplatin 100 mg m-2 intravenously at the beginning of each cycle, plus oral capecitabine 850 mg m-2 twice daily on days 1-14 of each cycle.

SUMMARY:
The investigators will conduct a prospective phase 2 study to evaluate the efficacy and safety of a modified neoadjuvant immunotherapy plus chemotherapy (one cycle of Tislelizumab monotherapy followed by four cycles of Tislelizumab plus Docetaxel, Oxaliplatin and Capecitabine) in patients with locally advanced resectable adenocarcinoma of the esophagogastric junction (AEG).

DETAILED DESCRIPTION:
Adenocarcinoma of the esophagogastric junction (AEG) has recently garnered increasing attention as a distinct type of malignancy. The World Health Organization (WHO) defines AEG as adenocarcinoma with its center located within 5 cm above or below the esophagogastric junction, crossing or abutting this junction (PMID: 31433515). Surgery remains the primary treatment for locally advanced AEG, but numerous studies have demonstrated that multimodal therapies, such as neoadjuvant chemoradiotherapy and chemotherapy, can achieve better outcomes.

The CROSS study (PMID: 22646630) established neoadjuvant chemoradiotherapy as the standard treatment for resectable esophageal and esophagogastric junction cancers. This trimodal approach not only significantly increased the R0 resection rate but also improved overall survival (OS). The FLOT4 study (PMID: 30982686) compared the efficacy and safety of perioperative FLOT chemotherapy with perioperative ECF chemotherapy in treating gastric cancer/AEG. The study found that the R0 resection rate was significantly higher in the FLOT group compared to the ECF/ECX group (85% vs. 78%). Patients in the FLOT group had a median OS of 50 months, compared to 35 months in the ECX/ECF group, demonstrating that intensified perioperative systemic therapy enhances neoadjuvant efficacy. Despite these advances, the overall prognosis for locally advanced AEG remains poor, with a 5-year survival rate of less than 45%. Thus, there is an urgent need for new treatment strategies to further improve perioperative chemotherapy outcomes for AEG.

Currently, immunotherapy combined with chemotherapy has become the first-line standard treatment recommendation for advanced esophageal cancer/AEG (CheckMate649, PMID: 34102137; Rationale 305, PMID: 38806195). In exploring perioperative immunotherapy for AEG, results from two global Phase III randomized controlled trials (KEYNOTE-585 (PMID: 38134948) and MATTERHORN (2023 ESMO. Abstract #LBA73)) indicated that neoadjuvant immunotherapy combined with chemotherapy significantly increased the pathological complete response rate (pCR) in AEG patients compared to neoadjuvant chemotherapy alone (13% vs. 2% and 17% vs. 7%, respectively). Furthermore, the neoadjuvant immunotherapy combined with chemotherapy groups did not show an increase in adverse events during the neoadjuvant period compared to the neoadjuvant chemotherapy alone groups (64% vs. 63% and 58% vs. 56%, respectively). However, the improvement in overall survival prognosis remains insufficient, suggesting the need to further optimize neoadjuvant immunotherapy protocols to achieve better therapeutic benefits.

The way for optimizing the treatment strategy for immune-chemotherapy includes the modifications of dose, drug selection, number of cycles, schedule and sequencing (PMID: 33712487). The PANDA study, initiated by Dutch researchers, is a single-arm Phase II clinical trial that enrolled 21 patients with resectable AEG (PMID: 38191613). The neoadjuvant treatment involved one induction cycle of single-agent immunotherapy (atezolizumab) followed by four cycles of sequential immunotherapy combined with DOC chemotherapy before surgery. The postoperative pCR rate was 45%, and the major pathological response (MPR) rate was 70% (13 out of 14 MPR patients achieved disease-free survival for up to four years). This study demonstrated that the initial induction with single-agent immunotherapy significantly altered the tumor immune microenvironment, inducing an immune activation state that provided a critical foundation for the efficacy of subsequent sequential immunotherapy combined with chemotherapy. The results suggest that an initial induction with single-agent immunotherapy prior to immunotherapy combining chemotherapy is a superior neoadjuvant immuno-chemotherapy strategy for resectable locally advanced AEG, warranting further exploration and validation in larger cohorts of AEG patients.

However, for Asia, particularly China, given the large base of esophageal cancer cases and the rising incidence of esophageal adenocarcinoma, exploring optimal neoadjuvant treatment strategies for resectable AEG patients in China has become a critical clinical issue.

This study aims to investigate the efficacy and safety of neoadjuvant immunotherapy induction followed by sequential immune-chemotherapy in patients with locally advanced AEG.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects signed the informed consent and volunteered to participate in the study.
2. Primary resectable, histologically confirmed Adenocarcinoma of the Esophagogastric junction (clinical stage T1-T4aN1-3M0 or T3-T4aN0M0, AJCC 8th).
3. Expect to have R0 resection
4. Age 18 or older.
5. ECOG PS: 0~1.
6. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, etc.
7. No contraindications to surgery.
8. Has sufficient organ function.
9. Women of childbearing age must undergo a serological pregnancy test within 7 days before first administration. Women of childbearing age, or male subjects with childbearing age female partners, must take contraceptive measures from the first dose to six months after last administration.
10. Good compliance, willing to comply with follow-up schedules.

Exclusion Criteria:

1. Subjects have received or are receiving any of:

1. anti-tumor interventions such as radiotherapy, chemotherapy, immunotherapy or other medications.
2. Received systemic corticosteroid therapy (prednisone equivalence> 10mg/d) or other immunosuppressive agents within the first 2 weeks prior to the first administration.
3. live vaccine within 4 weeks before the first administration.

2. Cancer related exclusion criteria:

1. other cancers instead of AEG
2. non-resectable or metastatic AEG
3. Subjects with other malignant tumors within 5 years before the first administration, but subjects with cervical carcinoma in situ, skin basal cell carcinoma, skin squamous cell carcinoma, and localized prostate cancer received radical surgery in situ that have received radical treatment and do not need other treatment can be included.

3. Other criteria: Subjects have uncontrolled cardiovascular diseases, such as 1) heart failure ≥ NYHA class 2, 2) unstable angina 3) myocardial infarction within 1 year; 4) supraventricular or ventricular arrythmia that needs treatment Subjects with any known active autoimmune disease Pregnant or breastfeeding female Presence of allergy or hypersensitivity to investigational medications HIV positive or active hepatitis B (HbsAg positive and HBV-DNA ≥2000 IU/ml or ≥ 104 copies/mL) or active hepatitis C (HCV antibody positive) or active tuberculosis Investigators assessed there might be other factors that cause subjects to withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06-19 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Through the study completion, an average of 12 months
  The primary endpoint is a pCR rate, which is defined as the absence of any remaining tumor cells in both the main tumor and the nearby lymph nodes (ypT0N0) as per the AJCC 8th Edition TRG scoring system

SECONDARY OUTCOMES:
MPR rate | Through the study completion, an average of 12 months
  The primary endpoint is a pCR rate, which is defined as the absence of any remaining tumor cells in both the main tumor and the nearby lymph nodes (ypT0N0) as per the AJCC 8th Edition TRG scoring system
Event-free survival (EFS) | Through the study completion, an average of 36 months
  An event-free survival (EFS) is defined as the duration from the start of treatment until disease progression/recurrence or death from any cause, whichever occurs first
Overall survival (OS) | Through the study completion, an average of 36 months
  Overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence
Adverse events and treatment-related adverse events | Through the study completion, an average of 12 months
  Including adverse events and complications. Incidence of adverse events using CTCAE 5.0; grade 3 treatment-related adverse events and higher-grade will be reported
R0 resection rate | Through the study completion, an average of 12 months
  A R0 resection rate is defined as the rate of complete tumor removal with negative resection margin microscopically
2-year recurrence-free survival between patients with postoperative ctDNA negative and postoperative ctDNA positive | From the completion of surgery to the completion of the 2-year postoperative follow-up.
  patients will have ctDNA detection at 2-4 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagtegaal ID, Odze RD, Klimstra D, Paradis V, Rugge M, Schirmacher P, Washington KM, Carneiro F, Cree IA; WHO Classification of Tumours Editorial Board. The 2019 WHO classification of tumours of the digestive system. Histopathology. 2020 Jan;76(2):182-188. doi: 10.1111/his.13975. Epub 2019 Nov 13. No abstract available. PMID 31433515
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Al-Batran SE, Homann N, Pauligk C, Goetze TO, Meiler J, Kasper S, Kopp HG, Mayer F, Haag GM, Luley K, Lindig U, Schmiegel W, Pohl M, Stoehlmacher J, Folprecht G, Probst S, Prasnikar N, Fischbach W, Mahlberg R, Trojan J, Koenigsmann M, Martens UM, Thuss-Patience P, Egger M, Block A, Heinemann V, Illerhaus G, Moehler M, Schenk M, Kullmann F, Behringer DM, Heike M, Pink D, Teschendorf C, Lohr C, Bernhard H, Schuch G, Rethwisch V, von Weikersthal LF, Hartmann JT, Kneba M, Daum S, Schulmann K, Weniger J, Belle S, Gaiser T, Oduncu FS, Guntner M, Hozaeel W, Reichart A, Jager E, Kraus T, Monig S, Bechstein WO, Schuler M, Schmalenberg H, Hofheinz RD; FLOT4-AIO Investigators. Perioperative chemotherapy with fluorouracil plus leucovorin, oxaliplatin, and docetaxel versus fluorouracil or capecitabine plus cisplatin and epirubicin for locally advanced, resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4): a randomised, phase 2/3 trial. Lancet. 2019 May 11;393(10184):1948-1957. doi: 10.1016/S0140-6736(18)32557-1. Epub 2019 Apr 11. PMID 30982686
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Qiu MZ, Oh DY, Kato K, Arkenau T, Tabernero J, Correa MC, Zimina AV, Bai Y, Shi J, Lee KW, Wang J, Poddubskaya E, Pan H, Rha SY, Zhang R, Hirano H, Spigel D, Yamaguchi K, Chao Y, Wyrwicz L, Disel U, Cid RP, Fornaro L, Evesque L, Wang H, Xu Y, Li J, Sheng T, Yang S, Li L, Moehler M, Xu RH; RATIONALE-305 Investigators. Tislelizumab plus chemotherapy versus placebo plus chemotherapy as first line treatment for advanced gastric or gastro-oesophageal junction adenocarcinoma: RATIONALE-305 randomised, double blind, phase 3 trial. BMJ. 2024 May 28;385:e078876. doi: 10.1136/bmj-2023-078876. PMID 38806195
- [Background] Shitara K, Rha SY, Wyrwicz LS, Oshima T, Karaseva N, Osipov M, Yasui H, Yabusaki H, Afanasyev S, Park YK, Al-Batran SE, Yoshikawa T, Yanez P, Dib Bartolomeo M, Lonardi S, Tabernero J, Van Cutsem E, Janjigian YY, Oh DY, Xu J, Fang X, Shih CS, Bhagia P, Bang YJ; KEYNOTE-585 investigators. Neoadjuvant and adjuvant pembrolizumab plus chemotherapy in locally advanced gastric or gastro-oesophageal cancer (KEYNOTE-585): an interim analysis of the multicentre, double-blind, randomised phase 3 study. Lancet Oncol. 2024 Feb;25(2):212-224. doi: 10.1016/S1470-2045(23)00541-7. Epub 2023 Dec 19. PMID 38134948
- [Background] Salas-Benito D, Perez-Gracia JL, Ponz-Sarvise M, Rodriguez-Ruiz ME, Martinez-Forero I, Castanon E, Lopez-Picazo JM, Sanmamed MF, Melero I. Paradigms on Immunotherapy Combinations with Chemotherapy. Cancer Discov. 2021 Jun;11(6):1353-1367. doi: 10.1158/2159-8290.CD-20-1312. Epub 2021 Mar 12. PMID 33712487
- [Background] Verschoor YL, van de Haar J, van den Berg JG, van Sandick JW, Kodach LL, van Dieren JM, Balduzzi S, Grootscholten C, IJsselsteijn ME, Veenhof AAFA, Hartemink KJ, Vollebergh MA, Jurdi A, Sharma S, Spickard E, Owers EC, Bartels-Rutten A, den Hartog P, de Miranda NFCC, van Leerdam ME, Haanen JBAG, Schumacher TN, Voest EE, Chalabi M. Neoadjuvant atezolizumab plus chemotherapy in gastric and gastroesophageal junction adenocarcinoma: the phase 2 PANDA trial. Nat Med. 2024 Feb;30(2):519-530. doi: 10.1038/s41591-023-02758-x. Epub 2024 Jan 8. PMID 38191613